CLINICAL TRIAL: NCT03606811
Title: The Role of Double Modality " Fluoroscopic &Ultrasonographic " Guidance of Superior Hypogastric Plexus Neurolysis in Treating Intractable Pelvic Cancer Pain: a Comparative Study.
Brief Title: Fluoroscopic &Ultrasonographic Guidance of Superior Hypogastric Plexus Neurolysis in Intractable Pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed H Othman, Assisstant professor of Anesthesia ICU and pain Relief, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IORG0003301
Record Dates: First submitted 2018-07-14; First posted 2018-07-31 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Intractable Pelvic Cancer Pain
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fluroscopic guided block (Active Comparator)
  Interventions: Procedure: fluroscopic guided block
- double modality guided block (Experimental)
  Interventions: Procedure: double modality (ultrasound and fluroscopic) guided block

INTERVENTIONS:
Procedure: fluroscopic guided block — SHPB will be done Fluoroscopic-guided (the posterior oblique trajectory technique.
  Arms: fluroscopic guided block
Procedure: double modality (ultrasound and fluroscopic) guided block — SHPB will be done using our described new technique of performing the modified Mishra technique by injecting 3-5 ml of contrast media (lohexol=omnipaque) after getting the target position. Then C-arm pictures will be checked (both P-A & dead lateral)
  Arms: double modality guided block

SUMMARY:
fluoroscopic group & includes 30 patients where SHPB will be done Fluoroscopic-guided (the posterior oblique trajectory technique.the double modality group & includes 30 patients where SHPB will be done using our described new technique of performing the modified Mishra technique by injecting 3-5 ml of contrast media (lohexol=omnipaque) after getting the target position.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Intractable pelvic cancer pain (VAS > 40 mm)
* Pain is refractory to pharmacotherapy (both opioids and adjuvant therapy) or opioids' side effects are not tolerated.

Exclusion criteria

* Local or systemic sepsis.
* Uncorrectable coagulopathy.
* Neuropsychiatric illness.
* History of drug abuse.
* Pregnant or lactating patients.
* Distorted local anatomy.
* Patients who are known to be allergic to the used medications.
* Cardiovascular or respiratory instability.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-05 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
pain relief will be assessed by VAS | 12 weeks
  pain relief will be assessed by VAS (visual Analogue score) which is 100 mscale with left (0) end means no pain & right (10) end means the worst possible pain

CONTACTS AND LOCATIONS:
Locations (1):
- NCI, Cairo university, Cairo, Egypt